CLINICAL TRIAL: NCT05869214
Title: Middle East African Registry Women CardioVascular Disease
Acronym: MEA-WCVD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tunisian Society of Cardiology and Cardiovascular Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: WCVD012023
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure; Atrial Fibrillation; Valvular Heart Disease; Ischemic Heart Disease
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation; Heart Valve Diseases; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MEA cardiology societies have joined forces to tackle the issue by establishing a tangible real-world data registry in every MEA country. This endeavor has resulted in the development of a multicenter registry called MEA-WCVD, which is being sponsored by each national cardiology society from participating countries. All data gathered will be consolidated into a singular registry for thorough analysis. Country specific analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* All incomers in Cardiovascular (CV) diseases in hospital or out hospital facilities with one of the 4 diagnosis (Heart Failure (HF), Atrial fibrillation (AF), Valvular Heart disease (VHD), ischemic heart disease (IHD)
* Age over 18 years old
* Men and Women
* Signature of consent form

Exclusion Criteria:

Patients with diseases other than the 4 previously mentioned in inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients having their consultation in the study participating site.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-07-10 (Estimated); Study Completion 2023-07-10 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular diseases care management in women will be compared to men in MEA countries according to current practice guidelines | 2 months

SECONDARY OUTCOMES:
Identify inequalities between both genders in terms of: • Healthcare insurance • Incomes • Access to healthcare | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hedi chaker Hospital, Sfax, Tunisia

IPD SHARING:
Plan to Share IPD: No